CLINICAL TRIAL: NCT03588169
Title: Representations of Oral Nutritional Supplementation (ONS) in Hospitals : Gender differences_observational Study
Acronym: CNO_ALIMS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BRINDISI 2018 CNO_ALIMS
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Malnutrition; Oral Nutritional Supplementation
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients hospitalized at the Dijon University Hospital: Patients hospitalized in the endocrinology, digestive surgery, pneumology and geriatric units of the Dijon University Hospital with a prescription for ONS
  Interventions: Dietary Supplement: semi-structured interviews

INTERVENTIONS:
Dietary Supplement: semi-structured interviews — About 30 minutes and touching on the following subjects:
  * perception of hospital meals
  * patient representation of ONS
  * taking ONS and feelings about it

SUMMARY:
Over 30% of hospitalized patients are malnourished. These figures range from 20% to 60% in geriatric units. Undernutrition results either from a decrease in energy intake, an increase in needs, an increase in losses or a combination of these three causes. As a factor in mortality, morbidity and lengthening the time of hospital stays, undernutrition induces health costs 45 to 102% higher than a person who is not undernourished. The nutritional management of patients initially includes hygieno-dietary advice, then the implementation of an oral nutritional supplementation (ONS). A recent study conducted by our teams highlighted the low ONS consumption among women compared to men (39.48% vs 73.41%). Interviews with patients showed that 13 out of 17 had a negative opinion of ONS.

The aim of this study is to show, on a larger scale, whether ONS consumption differs according to sex and if so, to highlight the obstacles to this consumption through the implementation of semi-directive interviews with patients. Ultimately, this research will lead to the implementation of alternative strategies to improve ONS consumption and to a better understanding of the obstacles to ONS consumption.

ELIGIBILITY:
Inclusion Criteria:

* patient who has given oral consent
* over 18 years
* orally fed
* with a prescription for ONS
* speaks and understands French
* hospital stay longer than 4 days

Exclusion Criteria:

* adult under tutelage
* pregnant or breastfeeding women
* cognitive disorders
* patient does not speak or understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised in the endocrinology, digestive surgery, pneumology and geriatrics departments of the Dijon University Hospital, with a prescription for ONS
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Semi-structured individual interviews | 1 day on inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France